CLINICAL TRIAL: NCT01293630
Title: An Open-label, Dose-escalation, Safety and Pharmacokinetics Phase I Study of Ombrabulin in Combination With Paclitaxel and Carboplatin Every 3 Weeks in Patients With Advanced Solid Tumors
Brief Title: A Dose-escalation Study of Ombrabulin in Combination With Paclitaxel and Carboplatin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD11270; U1111-1115-2568 (Other: UTN)
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — AC 7700; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort - 1 through 5 (Experimental): AVE8062 combined with paclitaxel and carboplatin will be administered once every 3 weeks
  Interventions: Drug: Ombrabulin (AVE8062); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Ombrabulin (AVE8062) — Pharmaceutical form:solution
  Route of administration: intravenous
Drug: Paclitaxel — Pharmaceutical form:solution
  Route of administration: intravenous
Drug: Carboplatin — Pharmaceutical form:solution
  Route of administration: intravenous

SUMMARY:
The primary objective of the study is to determine the maximum tolerated dose (MTD) based on the incidence of dose limiting toxicity (DLT) and the maximum administered dose (MAD) of ombrabulin combined with paclitaxel and carboplatin administered every 3 weeks in patients with advanced solid tumors.

Secondary Objectives:

* To assess the overall safety profiles of the combination therapy
* To characterize the pharmacokinetic profile of ombrabulin, its active metabolite RPR 258063, paclitaxel, and carboplatin when used in combination
* To document the objective tumor response

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 4-week screening phase, 21-day study treatment cycles, an end of treatment visit and a follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Patients with advanced solid tumor for which the combination paclitaxel and carboplatin is potentially effective such as lung cancer, epithelial ovarian cancer.
* Patients who have signed and dated an Institutional Review Board (IRB)-approved patient informed consent form prior to study enrollment or performance of any study-specific procedures.

Exclusion criteria:

* Less than 20 or above 75 years of age ECOG performance status ≥2.
* Patients with more than 1 line of previous chemotherapy for advanced or metastatic disease (adjuvant/neoadjuvant and targeted agents [eg gefitinib] excluded)
* Concurrent treatment with any other anticancer therapy (except palliative radiotherapy),
* Women of childbearing potential who does not agree with contraception.
* Washout period of less than 28 days from prior anticancer therapies
* Symptomatic brain metastases and carcinomatous leptomeningitis.
* Other serious illness or medical conditions
* Current peripheral neuropathy ≥grade 2 and ototoxicity,
* Absolute neutrophils counts<1.5 x 10E9/L. - Platelets count<100 x 10E9/L. - hemoglobin <9.0 g/dL (without red blood cell transfusion within 28 days before the test). - Creatinine Clearance<55 mL/min. - Total bilirubin >upper normal limits of the institutional norms. - ALT/AST >1.5 times the upper normal limits of the institutional norms. - AP>2.5 times the upper normal limits of the institutional norms.
* Medical history of myocardial infarction, angina pectoris, congestive heart failure, coronary artery bypass graft , arrhythmia , stroke or history of arterial or venous thrombo-embolism within the past 180 days requiring anticoagulants.
* Patient with a LVEF <50% by echocardiography.
* Patient with uncontrolled hypertension and patient with organ damage related to hypertension such as left ventricular hypertrophy or grade 2 ocular fundoscopic changes or kidney impairment.
* Hypertension defined as systolic BP >140 mmHg or diastolic BP >90 mmHg on two repeated measurements at 30 minutes interval.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The number of of drug related adverse events meeting the defined dose limiting toxicity at Cycle 1 | 3 weeks

SECONDARY OUTCOMES:
The number of treatment emergent adverse events | 30 days after the last injection
The number of serious adverse events | 30 days after the last injection
The number of laboratory abnormalities | 30 days after the last injection
Pharmacokinetic parameter of ombrabulin: Cmax | Day 1-2 at Cycle 1
Pharmacokinetic parameter of RPR258063: tmax | Day 1-2 at Cycle 1
Pharmacokinetic parameter of paclitaxel: Cmax | Day 1-3 at Cycle 1
Pharmacokinetic parameter of carboplatin (free and total platinum): Cmax | Day 1-3 at Cycle 1
Investigator determination of response | 30 days after the last injection
Pharmacokinetic parameter of ombrabulin: AUC | Day 1-2 at Cycle 1
Pharmacokinetic parameter of ombrabulin: CL | Day 1-2 at Cycle 1
Pharmacokinetic parameter of ombrabulin: Vss | Day 1-2 at Cycle 1
Pharmacokinetic parameter of ombrabulin: t 1/2 | Day 1-2 at Cycle 1
Pharmacokinetic parameter of RPR258063: Cmax | Day 1-2 at Cycle 1
Pharmacokinetic parameter of RPR258063: AUC | Day 1-2 at Cycle 1
Pharmacokinetic parameter of RPR258063: t 1/2 | Day 1-2 at Cycle 1
Pharmacokinetic parameter of RPR258063: Metabolic Ratio | Day 1-2 at Cycle 1
Pharmacokinetic parameter of paclitaxel: AUC | Day 1-3 at Cycle 1
Pharmacokinetic parameter of paclitaxel: CL | Day 1-3 at Cycle 1
Pharmacokinetic parameter of paclitaxel: Vss | Day 1-3 at Cycle 1
Pharmacokinetic parameter of paclitaxel: t 1/2 | Day 1-3 at Cycle 1
Pharmacokinetic parameter of carboplatin (free and total platinum): AUC | Day 1-3 at Cycle 1
Pharmacokinetic parameter of carboplatin (free and total platinum): CL | Day 1-3 at Cycle 1
Pharmacokinetic parameter of carboplatin (free and total platinum): Vss | Day 1-3 at Cycle 1
Pharmacokinetic parameter of carboplatin (free and total platinum): t 1/2 | Day 1-3 at Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Japan (2):
  - Investigational Site Number 392002, Akashi-Shi
  - Investigational Site Number 392001, Hidaka-Shi

REFERENCES:
- [Derived] Matsumoto K, Sunaga Y, Ecstein-Fraisse E, Fujiwara K. Phase I study of ombrabulin in combination with paclitaxel and carboplatin in Japanese patients with advanced solid tumors. Int J Gynecol Cancer. 2024 Apr 1;34(4):586-593. doi: 10.1136/ijgc-2022-003880. PMID 37989482